CLINICAL TRIAL: NCT02803476
Title: Is There An Association Between Vitamin D Levels And Insulin Resistance In Polycystic Ovary Syndrome?
Brief Title: Is There Association Between Vitamin D Levels And Insulin Resistance In Polycystic Ovary Syndrome?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Sara Saad Youssef Morsi, MD, Ain Shams Maternity Hospital
Other Study IDs: 2732016
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance; Vitamin D Deficiency
Keywords: PCO; Vitamin D; Insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Overnight fasting venous blood samples will be withdrawn between the 2nd and 3rd day of menstruation, and withdrawal bleeding following progesterone therapy for 5 days in amenorheic women, centrifuged and frozen to -80 C until analyzed for the assessment of vitamin D levels, Androgen levels, plasma Glucose and plasma Insulin, FSH and LH analogues.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: Polycystic ovary syndrome (PCOS) female patients. 20-35 years of age.
- Controls: Non-PCOs female subjects. 20-35 years of age.

SUMMARY:
The primary aim of the current study is to clarify whether serum vitamin D levels [25(OH)D3] have a temporal association with insulin resistance and/or insulin sensitivity in PCOS women versus healthy ones.

To achieve this aim, the investigators will conduct a prospective observational study involving obese and lean PCOS women in comparison to obese and lean healthy subjects living in Cairo, Egypt.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common gynecological endocrinopathy among women of reproductive age. The prevalence of PCOS among such women is estimated to be 6.4% to 6.8% worldwide. PCOS is a heterogeneous androgen excess disorder with different degrees of reproductive and metabolic dysfunctions.

There are many considerations to explain the complexity of the underlying pathogenesis of PCOS, particularly the well-known roles of hypothalamic-pituitary gonadal dysfunctions, metabolic abnormalities and genetic factors, the developmental model of chronic diseases postulates that early-life events affect the individual differences in vulnerability to lifestyle and environment, suggesting that hostile intrauterine environment and low birth weight may predispose to the development of early adrenarche, PCOS and metabolic syndrome later in life; however, the definite pathogenesis and real underlying etiologies of PCOS remain uncertain and ripe with opportunities for further research.

PCOS is the most common cause of anovulatory infertility, and its foremost clinical symptoms include anovulation or oligo-ovulation, infertility, menstrual irregularity, polycystic ovaries, and hyperandrogenism in women without specific underlying diseases of the adrenal or pituitary glands. A primary abnormality in folliculogenesis may have played a role in the development of PCOS. The polycystic ovaries contain multiple antral follicles, some of which prematurely acquire LH receptors and become responsive to LH, increasing granulosa cell proliferation in the preantral follicles, resulting in anovulation. PCOS is defined by the presence of having at least 2 of the following criteria: irregular or absent ovulation, elevated levels of androgenic hormones, and enlarged ovaries containing at least 12 follicles each.

Several epidemiological and interventional PCOS studies demonstrate that serum vitamin D concentrations are inversely associated with fasting plasma glucose levels, insulin resistance, body mass index (BMI), and body fat contributing to the pathogenesis of PCOS by promoting insulin resistance and affecting glucose metabolism in PCOS women. Vitamin D is either produced in the skin in response to direct exposure to sunlight from dehydrocholesterol or obtained from the diet. Vitamin D3 (cholecalciferol) is converted into 25-hydroxyvitamin D3 principally in the liver and 1,25-dihydroxyvitamin D3 in the kidney by two hydroxylation steps. 1,25-dihydroxyvitamin D3 is an active form of vitamin D, it binds to vitamin D receptors (VDRs) that are expressed in 2776 genomic positions and modulate the expression of 229 genes in more than 30 different tissues, such as the skeleton, pancreatic islet cells, parathyroid glands, and ovaries.

About 3% of the human genome are regulated by VDRs gene including those responsible for glucose and fat metabolism as well as blood regulation; it's active form acts through its VDRs either directly or through regulation of intercellular calcium that facilitates insulin secretion. It has been suggested that Vitamin D increases insulin sensitivity through the effect on its muscle cell receptors by increasing insulin receptors or increasing the insulin sensitivity of insulin receptors to insulin. Also, being a fat soluble vitamin, a higher proportion of vitamin D may be sequestered in the adipose tissue of obese individuals, resulting in lower 25-(OH)D3 concentration levels; therefore, a low vitamin D status is suspected to be a risk factor for impaired glucose tolerance, insulin resistance and a substantial cause of obesity.

In the light of the literature, the relationship between vitamin D status and insulin or glucose metabolism has been investigated in women with PCOS who are vitamin D deficient, although there is no consensus on whether or not serum vitamin D levels are different in women with or without PCOS. Vitamin D level is defined as a serum level of 25-hydroxycholecalciferol [25-(OH)D3]. Vitamin D insufficiency is defined as a 25-(OH)D3 concentration of <30ng/ml and frank vitamin D deficiency is defined as a 25-(OH)D3 concentration of <20ng/ml. There appears to be a growing disconnect between the observational studies and the randomized clinical trials of vitamin D supplementation in PCOS women with insulin resistance and glucose intolerance. Observational studies keep showing a fairly consistent relationship between low concentration levels of vitamin D and insulin resistance or glucose intolerance, while almost all randomized trials, including a meta-analysis of vitamin D supplementation on women suffering from PCOS shows minimal, if any, benefit in terms of correcting insulin resistance or increasing insulin sensitivity indexes or an improvement in glucose metabolism. The results published indicated that the change was not significant and did not show any difference in insulin resistance which is the core patho-physiology of this syndrome.

Vitamin D deficiency (VDD) is common in women with and without PCOS and may be associated with metabolic and endocrine disorders in PCOS. However, the phenotypic manifestation of PCOS is associated with various degrees of gonadotropic and/or metabolic abnormalities and there has been much debate as to whether it represents a single disorder or several that can only be determined by the interaction of multiple genetic and environmental factors. Previously conducted prospective observational studies that investigated the temporal relationship between VDD and metabolic disturbances (resistance to the action of insulin and glucose intolerance) in PCOS are lacking. If VDD were causally related to PCOS and the subsequent development of metabolic dysfunction in PCOS, then further prospective observational studies with repeated VDD assessment and better characterization of PCOS disease severity at enrollment are needed to clarify whether VDD is a co-determinant of metabolic dysregulations in PCOS compared to Non-PCOS women (controls).

Study design:

A prospective observational study which will be conducted in the outpatient clinics of Ain Shams University Women's Hospital after being approved by the local ethical committee.

Sample size justification:

For sample size determination, the investigators used the following formula: N= 2 x K x [SD/μ1-μ2]2 where N equals the number of patients per arm and K is constant (K=7.9) setting the type-1 error α at 0.5 and the power β at 80%. Results from a previous study calculated the mean (standard deviation (SD)) of vitamin Din the PCOS group(μ1)is 15.45 ± 7.88 ng/ml and in the control group(μ2) 12.83 ± 5.76ng/ml. Anticipating a 10% drop out rate, we calculated that a sample size of 83 subjects in each group, with a total of 166 subjects is enough to detect a significant difference, if any existed.

Objectives:

1. To measure plasma concentrations of vitamin D, fasting glucose, fasting Insulin, androgen levels, FSH and LH levels in all participants diagnosed with PCOS and healthy participants.
2. To clarify whether VDD is a co-determinant of metabolic dysregulations particularly insulin resistance and glucose metabolism in PCOS when compared to healthy women (controls).
3. To develop a better assessment of the PCOS severity and factors involved.

Methodology:

All of the recruited subjects will undergo:

* Written consent.
* Complete history with particular emphasis on menstrual, sexual, gynecological, medical as (Irregular cycles, oligomenorrhea, polymenorrhea, secondary amenorrhea, dysmenorrhea primary or secondary infertility, cancer, thyroid disease, galactorrhea, hirsutism, pelvic pain...etc), previous pelvic surgeries, induction of ovulation, vaginal infection, abnormal Pap smears, life style habits such as alcohol and smoking.
* Physical examination including general examination, Anthropometric measurements like weight (in kg), height (in meters), Body Mass Index (BMI), waist to hip ratio (WHR), Waist circumference (midway between the lowest rib margin and iliac crest) and hip circumference (over the widest part of the gluteal region). Signs of androgen excess, thyroid toxicity, and galactorrhea will be examined. Patients will undergo gynecological ultrasound in the follicular phase and to assess the ovarian size and morphology. Local examination to exclude uterine abnormalities, cervical tenderness, masses, vaginal infections and discharge.
* Diagnostic tests: Overnight fasting venous blood samples will be withdrawn between the 2nd and 3rd day of menstruation, and withdrawal bleeding following progesterone therapy for 5 days in amenorheic women, centrifuged and frozen to -80 C until analyzed for the assessment of vitamin D levels, Androgen levels, plasma Glucose and plasma Insulin, FSH and LH analogues.

All collected data will be tabulated and statistically analyzed.

Statistical analysis:

Descriptive statistics for measured variables will be expressed as range, mean and standard deviation (for metric data); range, median and interquartile range (for discrete data); and number and proportions (for categorical data).

Demographic data, primary and secondary outcomes of all women will be compared using t-test (for quantitative parametric measures), Mann-Whitney's U-test (for quantitative non-parametric measures) and chi-squared for Fisher's Exact tests (for categorical measures). Pearson's correlation coefficient (for metric variables) and Spearman's correlation coefficient (for rank variables) will be used to estimate association between variables. Microsoft Excel and SPSS for Windows will be used for data presentation and statistical analysis.

Ethical considerations:

The clinical research study will be conducted in accordance with the above mentioned design, safety and reporting of cases matching the relevant policies, requirements, and regulations of the Ethical Committee of the Department of Obstetrics and Gynecology - Faculty of Medicine, Ain Shams University Women's Hospital.

Consent procedure:

The investigator will make certain that an appropriate informed consent process is in place to ensure that potential research subjects, or their authorized representatives, are fully informed about the nature and objectives of the clinical study, the benefits of study participation and their rights as research subjects. The investigator will obtain a written, signed informed consent of each subject, or the subject's authorized representative, prior to performing any study-specific procedures on the subject. The investigator will retain the original signed informed consent form.

Subject confidentiality:

All evaluation forms, reports and other records that leave the site will not include unique personal data to maintain subject confidentiality.

ELIGIBILITY:
PCOS female patients criteria:

Inclusion Criteria:

* PCOS will be diagnosed in accordance with Rotterdam criteria.
* No relevant systemic diseases e.g. hypertension, DM.

Exclusion Criteria:

* Androgen secreting tumor.
* Cushing syndrome.
* Congenital adrenal hyperplasia.
* Hyperprolactinemia.
* Virilism.
* Pregnant or nursing.
* Conditions known to affect Vitamin D deficiency like renal disease, liver disease, gastrointestinal problems and malnutrition.
* Taking vitamin D or calcium supplements.
* Untreated hypothyroidism or hyperthyroidism.

Non-PCOS female subjects criteria:

* Regular menstrual cycles
* Not suffering from any conditions known to affect Vitamin D deficiency like renal disease, liver disease, gastro-Intestinal problems and malnutrition.
* Not taking vitamin D or calcium supplements.
* No relevant systemic diseases e.g. hypertension, DM.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this study, a total of 166 consenting women with and without PCOS will be asked to participate and divided into two groups; 83 female patients will represent PCOS recruited from the outpatient clinics of Ain Shams university maternity hospital, along with 83 non-PCOS women who will represent controls recruited after fulfilling specific criteria.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Quantitative Insulin Sensitivity Check Index (QUICKI) | After sample collection and analysis, through study completion, an average of 20 weeks.
  A validated measure of Insulin sensitivity based on fasting Insulin (uIU/mL) and Glucose (mg/dL).

SECONDARY OUTCOMES:
Fasting Plasma Insulin | 12 hours of fasting.
  Overnight fasting venous samples
Fasting Plasma Glucose | 12 hours of fasting.
  Overnight fasting venous samples.
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | After sample collection and analysis, through study completion, an average of 20 weeks.
  A validated measure of Insulin sensitivity based on fasting Insulin (uIU/mL) and Glucose (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Hisham M Fathi, Phd, MD, Study Chair — Professor of Obstetrics & Gynecology. Faculty of Medicine - Ain Shams University.; Sherif A Ashoush, Phd, MD, Study Director — Professor of Obstetrics & Gynecology. Faculty of Medicine - Ain Shams University.; Sara S Youssef, MD, Principal Investigator — MD, Obstetrics and Gynecology. Faculty of Medicine - Ain Shams University
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Abbasseya District., Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Yildizhan R, Kurdoglu M, Adali E, Kolusari A, Yildizhan B, Sahin HG, Kamaci M. Serum 25-hydroxyvitamin D concentrations in obese and non-obese women with polycystic ovary syndrome. Arch Gynecol Obstet. 2009 Oct;280(4):559-63. doi: 10.1007/s00404-009-0958-7. Epub 2009 Feb 13. PMID 19214546
- [Background] Boucher BJ, Mannan N, Noonan K, Hales CN, Evans SJ. Glucose intolerance and impairment of insulin secretion in relation to vitamin D deficiency in east London Asians. Diabetologia. 1995 Oct;38(10):1239-45. doi: 10.1007/BF00422375. PMID 8690178
- [Background] Orwoll E, Riddle M, Prince M. Effects of vitamin D on insulin and glucagon secretion in non-insulin-dependent diabetes mellitus. Am J Clin Nutr. 1994 May;59(5):1083-7. doi: 10.1093/ajcn/59.5.1083. PMID 8172095
- [Background] Thomson RL, Spedding S, Buckley JD. Vitamin D in the aetiology and management of polycystic ovary syndrome. Clin Endocrinol (Oxf). 2012 Sep;77(3):343-50. doi: 10.1111/j.1365-2265.2012.04434.x. PMID 22574874
- [Background] Dunaif A. Insulin resistance and the polycystic ovary syndrome: mechanism and implications for pathogenesis. Endocr Rev. 1997 Dec;18(6):774-800. doi: 10.1210/edrv.18.6.0318. PMID 9408743
- [Background] Selimoglu H, Duran C, Kiyici S, Ersoy C, Guclu M, Ozkaya G, Tuncel E, Erturk E, Imamoglu S. The effect of vitamin D replacement therapy on insulin resistance and androgen levels in women with polycystic ovary syndrome. J Endocrinol Invest. 2010 Apr;33(4):234-8. doi: 10.1007/BF03345785. Epub 2009 Oct 9. PMID 19820295
- [Background] Ardabili HR, Gargari BP, Farzadi L. Vitamin D supplementation has no effect on insulin resistance assessment in women with polycystic ovary syndrome and vitamin D deficiency. Nutr Res. 2012 Mar;32(3):195-201. doi: 10.1016/j.nutres.2012.02.001. PMID 22464806
- [Background] Lobo RA, Carmina E. The importance of diagnosing the polycystic ovary syndrome. Ann Intern Med. 2000 Jun 20;132(12):989-93. doi: 10.7326/0003-4819-132-12-200006200-00010. PMID 10858183
- [Background] Carmina E. Genetic and environmental aspect of polycystic ovary syndrome. J Endocrinol Invest. 2003 Nov;26(11):1151-9. doi: 10.1007/BF03345266. PMID 15008257
- [Background] Rosenfield RL. Clinical review: Identifying children at risk for polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Mar;92(3):787-96. doi: 10.1210/jc.2006-2012. Epub 2006 Dec 19. PMID 17179197
- [Result] Azziz R, Woods KS, Reyna R, Key TJ, Knochenhauer ES, Yildiz BO. The prevalence and features of the polycystic ovary syndrome in an unselected population. J Clin Endocrinol Metab. 2004 Jun;89(6):2745-9. doi: 10.1210/jc.2003-032046. PMID 15181052
- [Result] Gluckman PD, Hanson MA, Cooper C, Thornburg KL. Effect of in utero and early-life conditions on adult health and disease. N Engl J Med. 2008 Jul 3;359(1):61-73. doi: 10.1056/NEJMra0708473. No abstract available. PMID 18596274
- [Result] Barber TM, Dimitriadis GK, Andreou A, Franks S. Polycystic ovary syndrome: insight into pathogenesis and a common association with insulin resistance. Clin Med (Lond). 2016 Jun;16(3):262-6. doi: 10.7861/clinmedicine.16-3-262. PMID 27251917
- [Result] Franks S, Stark J, Hardy K. Follicle dynamics and anovulation in polycystic ovary syndrome. Hum Reprod Update. 2008 Jul-Aug;14(4):367-78. doi: 10.1093/humupd/dmn015. Epub 2008 May 22. PMID 18499708
- [Result] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Result] Wehr E, Pilz S, Schweighofer N, Giuliani A, Kopera D, Pieber TR, Obermayer-Pietsch B. Association of hypovitaminosis D with metabolic disturbances in polycystic ovary syndrome. Eur J Endocrinol. 2009 Oct;161(4):575-82. doi: 10.1530/EJE-09-0432. Epub 2009 Jul 23. PMID 19628650
- [Result] Hahn S, Haselhorst U, Tan S, Quadbeck B, Schmidt M, Roesler S, Kimmig R, Mann K, Janssen OE. Low serum 25-hydroxyvitamin D concentrations are associated with insulin resistance and obesity in women with polycystic ovary syndrome. Exp Clin Endocrinol Diabetes. 2006 Nov;114(10):577-83. doi: 10.1055/s-2006-948308. PMID 17177140
- [Result] Ramagopalan SV, Heger A, Berlanga AJ, Maugeri NJ, Lincoln MR, Burrell A, Handunnetthi L, Handel AE, Disanto G, Orton SM, Watson CT, Morahan JM, Giovannoni G, Ponting CP, Ebers GC, Knight JC. A ChIP-seq defined genome-wide map of vitamin D receptor binding: associations with disease and evolution. Genome Res. 2010 Oct;20(10):1352-60. doi: 10.1101/gr.107920.110. Epub 2010 Aug 24. PMID 20736230
- [Result] Kumar S, Davies M, Zakaria Y, Mawer EB, Gordon C, Olukoga AO, Boulton AJ. Improvement in glucose tolerance and beta-cell function in a patient with vitamin D deficiency during treatment with vitamin D. Postgrad Med J. 1994 Jun;70(824):440-3. doi: 10.1136/pgmj.70.824.440. PMID 8029165
- [Result] He C, Lin Z, Robb SW, Ezeamama AE. Serum Vitamin D Levels and Polycystic Ovary syndrome: A Systematic Review and Meta-Analysis. Nutrients. 2015 Jun 8;7(6):4555-77. doi: 10.3390/nu7064555. PMID 26061015
- [Result] Lin MW, Wu MH. The role of vitamin D in polycystic ovary syndrome. Indian J Med Res. 2015 Sep;142(3):238-40. doi: 10.4103/0971-5916.166527. No abstract available. PMID 26458338
- [Result] Pal L, Berry A, Coraluzzi L, Kustan E, Danton C, Shaw J, Taylor H. Therapeutic implications of vitamin D and calcium in overweight women with polycystic ovary syndrome. Gynecol Endocrinol. 2012 Dec;28(12):965-8. doi: 10.3109/09513590.2012.696753. Epub 2012 Jul 11. PMID 22780885
- [Result] Nestler JE, Reilly ER, Cheang KI, Bachmann LM, Downs RW Jr. A pilot study: effects of decreasing serum insulin with diazoxide on vitamin D levels in obese women with polycystic ovary syndrome. Trans Am Clin Climatol Assoc. 2012;123:209-19; discussion 219-20. PMID 23303986
- [Result] Raja-Khan N, Shah J, Stetter CM, Lott ME, Kunselman AR, Dodson WC, Legro RS. High-dose vitamin D supplementation and measures of insulin sensitivity in polycystic ovary syndrome: a randomized, controlled pilot trial. Fertil Steril. 2014 Jun;101(6):1740-6. doi: 10.1016/j.fertnstert.2014.02.021. Epub 2014 Mar 14. PMID 24636395
- [Result] Campbell MJ, Julious SA, Altman DG. Estimating sample sizes for binary, ordered categorical, and continuous outcomes in two group comparisons. BMJ. 1995 Oct 28;311(7013):1145-8. doi: 10.1136/bmj.311.7013.1145. PMID 7580713
- [Result] Cook JA, Hislop J, Adewuyi TE, Harrild K, Altman DG, Ramsay CR, Fraser C, Buckley B, Fayers P, Harvey I, Briggs AH, Norrie JD, Fergusson D, Ford I, Vale LD. Assessing methods to specify the target difference for a randomised controlled trial: DELTA (Difference ELicitation in TriAls) review. Health Technol Assess. 2014 May;18(28):v-vi, 1-175. doi: 10.3310/hta18280. PMID 24806703
- [Result] Fox N, Mathers N. Empowering research: statistical power in general practice research. Fam Pract. 1997 Aug;14(4):324-9. doi: 10.1093/fampra/14.4.324. PMID 9283855
- [Result] Nishida C, Ko GT, Kumanyika S. Body fat distribution and noncommunicable diseases in populations: overview of the 2008 WHO Expert Consultation on Waist Circumference and Waist-Hip Ratio. Eur J Clin Nutr. 2010 Jan;64(1):2-5. doi: 10.1038/ejcn.2009.139. Epub 2009 Nov 25. PMID 19935820
- [Result] Hollis BW. Assessment and interpretation of circulating 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D in the clinical environment. Endocrinol Metab Clin North Am. 2010 Jun;39(2):271-86, table of contents. doi: 10.1016/j.ecl.2010.02.012. PMID 20511051
- [Result] Johnstone EB, Rosen MP, Neril R, Trevithick D, Sternfeld B, Murphy R, Addauan-Andersen C, McConnell D, Pera RR, Cedars MI. The polycystic ovary post-rotterdam: a common, age-dependent finding in ovulatory women without metabolic significance. J Clin Endocrinol Metab. 2010 Nov;95(11):4965-72. doi: 10.1210/jc.2010-0202. Epub 2010 Aug 18. PMID 20719841
- [Result] Adams JS, Hewison M. Update in vitamin D. J Clin Endocrinol Metab. 2010 Feb;95(2):471-8. doi: 10.1210/jc.2009-1773. PMID 20133466